CLINICAL TRIAL: NCT03492359
Title: Tidal Breathing Patterns Measured by Thora-3DI™ Structured Light Plethysmography for Evaluation of Severity of Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Thora-3DI™ for Evaluation of Severity of Chronic Obstructive Pulmonary Disease (COPD)
Acronym: SLPCOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landon Pediatric Foundation (Other)
Collaborators: Pneumacare Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SLP CL1
Record Dates: First submitted 2017-07-05; First posted 2018-04-10 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, Structured Light Plethysmography, COPD severity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Plethysmography, Whole Body; Spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Normal Control (Active Comparator): Participants with no diagnosis of respiratory disease between the ages of 0 and 80 whose breathing will be measured using Thora-3Di structured light plethysmography, body plethysmography and spirometry.
  Interventions: Device: Thora-3Di; Device: Body Plethysmography; Device: Spirometry
- COPD Patients (Active Comparator): Participants with chronic obstructive pulmonary disease between the ages of 0 and 80 whose breathing will be measured using Thora-3Di structured light plethysmography, body plethysmography and spirometry.
  Interventions: Device: Thora-3Di; Device: Body Plethysmography; Device: Spirometry

INTERVENTIONS:
Device: Thora-3Di — Device that uses a grid of structured light to measure chest and abdominal wall movement
  Other Names: Structured Light Plethysmography
Device: Body Plethysmography — A pulmonary function test (PFT) for measuring total lung volume.
Device: Spirometry — A pulmonary function tests (PFT) for measuring maximal forced expiratory flow and volume.

SUMMARY:
To demonstrate differences in tidal breathing patterns measured by SLP(Structured Light Plethysmography) between healthy subjects and COPD (chronic obstructive pulmonary disease). The correlation between SLP parameters and standard lung function parameters measured by body box and spirometry will also be assessed. Trends in SLP breathing patterns between the different GOLD (Global Initiative for Chronic Obstructive Lung Disease) stages of COPD, and between those and healthy subjects, will be investigated to assess whether SLP can detect differences between groups.

DETAILED DESCRIPTION:
Structured light plethysmography (SLP) is a novel, non-contact method for assessing quiet 'tidal' breathing. A number of studies have reported the effects of conditions such as chronic obstructive pulmonary disease (COPD) on tidal breathing patterns, and a previous study has shown that SLP is able to detect differences in ten tidal breathing patterns between healthy subjects and patients with COPD. In this present study, the investigators will aim to confirm the previous findings and also to examine the relationship between SLP tidal breathing parameters and traditional measurements of lung function measured by spirometry and body box plethysmograph. The correlation between SLP parameters with lung Function parameters measured by spirometry and body box plethysmography: forced expiratory volume in one second (FEV1); Forced vital capacity (FVC), FEV1/FVC (forced expiratory volume in one second/forced vital capacity); total lung capacity (TLC) and residual volume (RV). Trends in tidal breathing patterns between varying severities of COPD (based on the (Global initiative for lung disease (GOLD) grading system.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-80 years,
* BMI range 18-40 kg/m2
* Patients diagnosed, or suspected, with COPD or normal subjects with no previous or current diagnosis of respiratory disease

Exclusion Criteria:

* Patient unable to sit in an upright position for required period of time
* Patients with significant co morbidities (assessed by the clinician at screening only):
* Significant unilateral lung disease e.g. pneumonectomy
* Chest wall or spinal deformity e.g. scoliosis
* Obstructive sleep apnea (OSA), Apnoea hypopnoea index > 30 (if known)
* BMI>40
* Inability to consent/comply with trial protocol
* Presence of an acute disease process that might interfere with test performance, e.g. Nausea, vomiting, persistent coughing)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Difference in SLP Breath Timing indices measured in seconds and between Patients and Healthy Subjects | Baseline
  SLP breathing parameters derived from the movement of the thoracoabdominal (TA) wall during tidal breathing
Difference in SLP derived Relative Contribution (measured in %) between Patients and Healthy Subjects | Baseline
  SLP breathing parameters derived from the movement of the thoracoabdominal (TA) wall during tidal breathing that describes the contribution of a region of the thoracoabdominal wall to total displacement
Difference in SLP derived Phase (measured in degrees) between Patients and Healthy Subjects | Baseline
  SLP breathing parameters derived from the movement of the thoracoabdominal (TA) wall during tidal breathing that describes the contribution of a region of the thoracoabdominal wall to total displacement
Difference in SLP derived displacement rate derived parameters (measured in distance per second) between Patients and Healthy Subjects | Baseline
  SLP breathing parameters derived from the trace of displacement rate over time of the thoracoabdominal (TA) wall during tidal breathing
Difference in SLP displacement rate derived ratios between Patients and Healthy Subjects (measured in distance per second) between Patients and Healthy Subjects | Baseline
  SLP breathing parameters ratios derived from the trace of displacement rate over time of the thoracoabdominal (TA) wall during tidal breathing
Correlation between SLP parameters with lung Function parameters measured by spirometry and body box plethysmography ( FEV1; FEV1/FVC; TLC and RV) | Baseline
  SLP breathing parameters ratios derived from the trace of displacement rate over time of the thoracoabdominal (TA) wall during tidal breathing correlated with lung function measured by body plethysmography and spirometry

SECONDARY OUTCOMES:
The trends in tidal breathing patterns between varying severities of COPD (based on the GOLD grading system). | Baseline
  The trends in tidal breathing patterns between varying severities of COPD as measured by the GOLD grading system.

CONTACTS AND LOCATIONS:
Locations (1):
- Ventura County Medical Center, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ghezzi M, Tenero L, Piazza M, Bodini A, Piacentini G. Structured light plethysmography: new method to evaluate expiratory flow limitation in asthmatic children. Eur Respir J. 2015;46(suppl 59):PA3641.
- [Background] Hmeidi H, Chadwick E, Lenney W, et al. IE50 measured by structured light plethysmography (SLP) can differentiate between children with and without asthma, and can detect response to a bronchodilator. Am J Respir Crit Care Med. 2016;193 Meeting Abstracts:A4505.
- [Background] Hmeidi H, Chadwick E, Lenney W, et al. Structured light plethysmography (SLP) can quantify abnormal breathing in children aged 2-12 admitted with acute asthma. Am J Respir Crit Care Med. 2016;193 Meeting Abstracts:A4506.
- [Background] Chen Y, Xin Z, Qin C. Analysis of tidal breathing flow-volume curves in stable COPD patients. Chinese J Prac Intern Med. 2005;11:978-980.
- [Background] Kostianev S, Hristova A, Iluchev D. Characteristics of tidal expiratory flow pattern in healthy people and patient with chronic obstructive pulmonary disease. Folia Med (Plovdiv). 1999;41(3):18-25. PMID 10658362
- [Background] Williams EM, Madgwick RG, Morris MJ. Tidal expired airflow patterns in adults with airway obstruction. Eur Respir J. 1998 Nov;12(5):1118-23. doi: 10.1183/09031936.98.12051118. PMID 9864007
- [Background] Stick S. Measurements during tidal breathing. In: Stocks J, Sly P, Tepper R, Morgan W, eds. Infant respiratory function testing: Wiley-Liss; 1996:117-138.
- [Background] Motamedi-Fakhr S, Wilson RC, Iles R. Tidal breathing patterns derived from structured light plethysmography in COPD patients compared with healthy subjects. Med Devices (Auckl). 2016 Dec 29;10:1-9. doi: 10.2147/MDER.S119868. eCollection 2017. PMID 28096696
- [Background] Poole KA, Thompson JR, Hallinan HM, Beardsmore CS. Respiratory inductance plethysmography in healthy infants: a comparison of three calibration methods. Eur Respir J. 2000 Dec;16(6):1084-90. doi: 10.1034/j.1399-3003.2000.16f11.x. PMID 11292110
- [Background] Parreira VF, Vieira DS, Myrrha MA, Pessoa IM, Lage SM, Britto RR. Optoelectronic plethysmography: a review of the literature. Rev Bras Fisioter. 2012 Nov-Dec;16(6):439-53. Epub 2012 Nov 27. English, Portuguese. PMID 23184278
- [Background] de Boer W, Lasenby J, Cameron J, Wareham R, Ahmad S, Roach C et al.SLP:a zero-contact non-invasive method for pulmonary function testing. In: Labrosse F, Zwiggelaar R, Liu Y, Tiddeman B (eds). Proceedings of the British Machine Vision Conference. Aberystwyth: BMVA Press, 2010, 85.1-12. Availble at http://www.bmva.o
- [Background] Whitley E, Ball J. Statistics review 4: sample size calculations. Crit Care. 2002 Aug;6(4):335-41. doi: 10.1186/cc1521. Epub 2002 May 10. PMID 12225610